CLINICAL TRIAL: NCT05589350
Title: Comparison of the Impact of Saturated Fat From High-fat Yogurt or Low-fat Yogurt and Butter on Cardiometabolic Risk Markers: a Randomized Cross-over Trial
Brief Title: High-fat Yogurt and Plasma Lipids Profile
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University (Other)
Responsible Party: Principal Investigator, Javad Nasrollahzadeh, Associate Professor, Shahid Beheshti University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 32333
Record Dates: First submitted 2022-10-15; First posted 2022-10-21 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Plasma Lipid Profile

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-fat yogurt (Experimental): Daily consumption of 1-2 servings (based on daily calorie requirement) of high-fat yogurt
  Interventions: Other: saturated fat intake
- Low-fat yogurt and butter (Active Comparator): Daily consumption of 1-2 servings of low-fat yogurt along with daily consumption of about 10 grams of animal butter
  Interventions: Other: saturated fat intake

INTERVENTIONS:
Other: saturated fat intake — Intake of saturated fat from yogurt and animal butter daily for 4-week period

SUMMARY:
The goal of this clinical trial is to compare the effect of saturated fat intake from different source on cardiometabolic risk markers in healthy subjects. The main question it aims to answer are:

-Does intake of saturated fat in the form of high-fat yogurt have a different effect on cardiometabolic risk factors than intake of the same amount from butter? In this study, in two periods of 4 weeks, the effect of receiving saturated fat from high-fat yogurt compared to receiving the same amount of saturated fat from butter and low-fat yogurt on the plasma concentration of lipids, cholesterol, insulin, and some inflammatory factors will be studied in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy people who do not use lipid-lowering, blood pressure control or diabetes medications

Exclusion Criteria:

* Taking supplements of omega-3 fatty acids, or antioxidants

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-10-15 (Actual); Primary Completion 2023-04-13 (Actual); Study Completion 2023-04-13 (Actual)

PRIMARY OUTCOMES:
Plasma lipid profile | 4 weeks
  Plasma concentrations of cholesterol, high-density lipoprotein cholesterol, Low-density lipoprotein cholesterol, and triglyceride

SECONDARY OUTCOMES:
Glycemic measures | 4 weeks
  Fasting plasma concentrations of glucose and insulin

OTHER OUTCOMES:
Inflammatory markers | 4 weeks
  Plasma concentrations of c-reactive protein and interleukin 6

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Nutrition Research Unit, National Nutrition and Food Technology Research Institute, Tehran, Iran

REFERENCES:
- [Derived] Ranjbar YR, Nasrollahzadeh J. Comparison of the impact of saturated fat from full-fat yogurt or low-fat yogurt and butter on cardiometabolic factors: a randomized cross-over trial. Eur J Nutr. 2024 Jun;63(4):1213-1224. doi: 10.1007/s00394-024-03352-8. Epub 2024 Feb 17. PMID 38367032